CLINICAL TRIAL: NCT06191003
Title: Analysis of Urdu Version of Maastricht Upper Extremity Questionnaire: A Reliability and Validity Study.
Brief Title: Urdu Version of Maastricht Upper Extremity Questionnaire Reliability Validity Study.
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC-FSD-00249
Record Dates: First submitted 2023-12-19; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-12

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study, the examiners will investigate the reliability and validity of Mastrict Upper Extremity scale in Urdu language in Pakistani patients with Carpal tunnel syndrome.

DETAILED DESCRIPTION:
The objective of this study is to translate as well as culturally adapt the Mastrict Upper Extrimity scale (MUEQ) into Urdu language and to test its reliability and validity in patients with Carpal Tunnel Syndrome. This cross-sectional survey will use convenience sampling technique to enroll the participants on a pre-defined criteria.

The outcomes of this study will help in finding the reliability and validity of MUEQ in patients with CTS. The reliability of this scale will be examined using internal consistency and test-retest methods. The internal consistency will be checked by Cronbach's alpha value. The test-retest reliability will be analyzed using an interclass correlation with patients.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who had to execute computer jobs in office.
* Individuals who have been working in present position for minimum 6 months
* Individuals who have been working for at least 4 hours or more in a day

Exclusion Criteria:

* Individuals who had Severe phsycytric and behavioral complaint
* Individuals who had prior injury of upper extremity
* Individuals who had any surgery of upper extremity

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pakistani computer user's population with complaint of arm, neck, shoulder (CANS) was included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-04-28 (Actual); Study Completion 2023-04-28 (Actual)

PRIMARY OUTCOMES:
Visual Analouge scale | 12th week
  The visual analogue scale is a simple and frequently used method for the assessment of variations in intensity of pain. In clinical practice the percentage of pain relief, assessed by Visual Analouge scale, is often considered as a measure of the efficacy of treatment.
JAMAR Hydraulic hand Dynamometer | 12th week
  Hand grip strength is an indicator of general muscle strength that is measured using a hand dynamometer.
Boston questionnaire | 12th week
  The Boston Carpal Tunnel Score is a patient-reported questionnaire that examines symptom severity and overall functional status of patients with carpal tunnel syndrome.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, Study Chair — Riphah International University
Locations (1):
- Riphah International University, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No